CLINICAL TRIAL: NCT05337618
Title: Improving Neurotrauma by Depolarization Inhibition With Combination Therapy (INDICT): a Phase 2 Randomized, Feasibility Trial
Brief Title: Improving Neurotrauma by Depolarization Inhibition With Combination Therapy (INDICT)
Acronym: INDICT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: University of New Mexico (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jed Hartings, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Not yet assigned
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two study groups based on a block design with randomized block sizes of 2, 4 or 6 determined individually for each study site.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SD-Guided Care (Experimental): In this arm, ECoG data will be reviewed for SDs in real-time using the bedside clinical CNS monitor. As a secondary measure, recognition of SDs will be facilitated by custom software on a laptop that receives data from the CNS monitor. Data on SD occurrence will be used to guide treatment in a tier-based therapeutic escalation and de-escalation protocol with the goal of SD suppression. Therapies to be used among the tiers include adjusted targets for MAP, CPP, PaCO2, plasma glucose, temperature, as well as ketamine pharmacotherapy. Changes between tiers are determined by the success or failure of SD suppression at the given treatment level.
  Interventions: Diagnostic Test: Full-band Electrocorticography; Combination Product: Treatment Algorithm
- Standard ICU Care (No Intervention): Management in the Standard ICU Care arm will follow published national guidelines consisting of common ICU-based targets for physiologic intervention that are thought to mitigate the development of secondary brain injuries.
  Continuous ECoG monitoring will be performed for seizure monitoring, but information on the course of SDs in these patients will not be used to guide care. To enforce blinding to SD-related ECoG data, the ECoG bedside software will be locked with password protection to prevent displays with frequency filtering and time/amplitude scales that are necessary to identify SDs.

INTERVENTIONS:
Diagnostic Test: Full-band Electrocorticography — Diagnosis of spreading depolarizations in continuous electrocorticography
  Arms: SD-Guided Care
Combination Product: Treatment Algorithm — Protocol for escalation and de-escalation of physiologic-targeted and pharmacologic therapies to treat and prevent spreading depolarizations
  Arms: SD-Guided Care

SUMMARY:
This study is a randomized Phase 2 trial to determine the feasibility of real-time electrocorticographic monitoring of spreading depolarizations (SD) to guide implementation of a tier-based protocol of intensive care therapies, aimed at SD suppression, for the management of patients who have undergone acute operative treatment of severe traumatic brain injury.

DETAILED DESCRIPTION:
The goal of acute TBI treatment is to minimize secondary damage that evolves over hours to days after the primary injury. Until now, however, there have been no methods for monitoring heterogeneous pathologic mechanisms to identify patients for appropriate neuroprotection therapies. Using invasive monitoring, investigators have documented that spreading depolarizations (SD), a cytotoxic dysfunction of cerebral gray matter that has been well-characterized through 60 years of research in animal models, are the dominant pathophysiologic process in peri-lesion cortex of many, but not all, severe TBI patients. Furthermore, it was found that the occurrence of SD as a secondary injury process in patients is an independent predictor of worse neurologic outcomes. Thus, monitoring of SD as a heterogeneous mechanism in TBI may allow selective use of therapy in only those patients who might benefit.

Here the investigators will conduct a randomized Phase 2 feasibility trial that uses real-time SD monitoring to guide implementation of a tier-based protocol of intensive care therapies aimed at SD suppression. The study is based on the hypothesis that outcomes from severe TBI can be improved by targeting intensive care therapies to suppress the pathology of SDs as a brain marker and mechanism of secondary injury. The objective of this study is to test the feasibility of this approach to intensive care management of severe TBI in a Phase 2 trial that uses real-time SD monitoring to guide administration of prescribed therapies to suppress SD. The aims are to (1) determine the feasibility of real-time SD monitoring to guide intensive care management of severe TBI, and (2) determine the effect of SD-guided vs. standard care management to reduce secondary brain insults in severe TBI.

This is a randomized Phase 2 clinical trial enrolling approximately 72 patients at 3 sites. Patients requiring neurological surgery for emergency treatment of TBI will be enrolled. The need for surgery allows for the placement of an electrode strip on the brain during surgery for subsequent electrocorticography (ECoG). ECoG data will be monitored continuously in real-time for the occurrence of SDs during intensive care. When SDs are observed, these patients (~60%, or n=43) will be randomized 1:1 to either standard (control) or SD-guided care. In the standard care arm, treatment will follow local and national guidelines with blinding to further ECoG results. In the SD-guided arm, treatment will follow a tiered-based protocol with escalation and de-escalation based on efficacy to suppress further SD pathology. Treatments will include use of ketamine sedation and adjusted targets for plasma glucose, cerebral perfusion pressure, temperature, and end-tidal CO2.

As outcomes, the accuracy of real-time SD scoring and compliance with protocol tier assignment and therapy implementation will be assessed. The burden of SD pathology, other measures of cerebral physiology (intracranial and cerebral perfusion pressures, and brain oxygenation), and medical complications will also be compared between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

(1) clinical indication for emergency craniotomy with dural opening to treat acute TBI within 72 hr post-trauma

Exclusion Criteria:

1. persistent bilateral non-reactive pupils or other evidence of non-survivable injury,
2. decompressive craniectomy to treat refractory ICP subsequent to diffuse injury, (3) co-enrollment in another therapeutic TBI trial, and

(4) pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Burden of spreading depolarizations | During the period of intensive care invasive monitoring, up to two weeks after injury
  Spreading depolarization events will be scored based on review of electrocorticographic recordings. The number of depolarizations per recording day over the period of monitoring will serve as the measure of total burden. The burdens computed for patients will be compared between the two randomization arms.

SECONDARY OUTCOMES:
Burden of elevated intracranial pressure | During the period of intensive care invasive monitoring, up to two weeks after injury
  The time integral of the continuously monitored intracranial pressure signal above 22 mmHg will be computed for each patient as the measure of burden. The burdens computed for patients will be compared between the two randomization arms.
Burden of cerebral hypoxia | During the period of intensive care invasive monitoring, up to two weeks after injury
  The time integral of the continuously monitored cerebral oxygenation below 20 mmHg will be computed for each patient as the measure of burden. The burdens computed for patients will be compared between the two randomization arms.
Burden of low cerebral perfusion | During the period of intensive care invasive monitoring, up to two weeks after injury
  The time integral of the continuously monitored cerebral perfusions pressure below 60 mmHg will be computed for each patient as the measure of burden. The burdens computed for patients will be compared between the two randomization arms.
Glasgow Outcome Score-Extended | 6 months post-injury
  Scores on the GOS-E will be compared between the two randomization arms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). Data will also be shared through the Federal Interagency Traumatic Brain Injury Registry (FITBIR).